CLINICAL TRIAL: NCT03392077
Title: The Role of Digital Cervical Opening in Elective Cesarean Section
Brief Title: Digital Cervical and Cesarean Section
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Lecturer, Assiut University
Other Study IDs: DCCS
Record Dates: First submitted 2018-01-02; First posted 2018-01-05 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Caesarean Section
MeSH Terms: interventions — Cesarean Section; Labor Stage, First

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: cervical dilatation: patients who will have cervical dilatation during Caesarean section
  Interventions: Procedure: Caesarean section; Other: cervical dilatation
- Group A: non cervical dilatation: patients who will have not cervical dilatation during Caesarean section
  Interventions: Procedure: Caesarean section; Other: No cervical dilatation

INTERVENTIONS:
Procedure: Caesarean section — Caesarean section will be done to deliver the baby
Other: cervical dilatation — Cervical dilatation will be done by double gloves digital dilatation postpartum
  Groups: Group A: cervical dilatation
Other: No cervical dilatation — after delivery of the baby cervix will be remain closed
  Groups: Group A: non cervical dilatation

SUMMARY:
Cesarean delivery is one of the most commonly performed surgical operations worldwide Cesarean delivery even as an elective procedure has been associated with considerable maternal risks compared with vaginal delivery. Some of the complications include postpartum hemorrhage, uterine infection, urinary tract infection, wound infection, septicemia and maternal death. Over the years, many variations in the surgical technique of Cesarean delivery have been employed with the main purpose of improving its safety. A woman's cervix is firm and undilated at the beginning of pregnancy, but progressive remodeling occurs during gestation until the cervix is soft at term, especially the nulliparous cervix . The progressive dilatation of the cervix needs uterine contraction during labor. A mechanical dilatation of the cervix at cesarean section is defined as an artificial dilatation of the cervix performed by finger, sponge forceps or other instruments at non-labor cesarean section. According to a cochrane view The information currently available about the advantages of cervical dilatation at cesarean section is inconclusive. This may be due to small sample sizes and low power of statistic.

ELIGIBILITY:
Inclusion Criteria:

1. All women scheduled for elective cesarean section will be approached.
2. Women accepted to participate in the study participation after discussing the nature of the study.

Exclusion Criteria:

1. Immuno-compromised women.
2. Women suffering from any coagulation disorder or Blood disease.
3. Blood transfusion during surgery or before it.
4. History of wound infection or endometritis .
5. Ante partum hemorrhage.
6. History of long corticosteroid use.
7. Women refuse to participate in the study.
8. Suspected clinical evidence of infection.
9. anemic women
10. Multiple pregnancy
11. Preterm births
12. Rupture of membranes or chorioamnionitis
13. Women who use antibiotics during the last 24 hours due to any infection but not prophylactic antibiotic during caesarian section
14. Emergency caesarean section

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: women who will subjected to elective Cesarean section
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
The amount of postpartum blood loss (ml) | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Woman's Health Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided